CLINICAL TRIAL: NCT05300243
Title: The Predictive Role of HPV Integration in HSIL and Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-S140
Record Dates: First submitted 2022-02-03; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2021-07

CONDITIONS: HPV Integration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HPV integration test — The stratified analysis by the level of HPV DNA integration in HSIL and cervical cancer will be drawn to explore whether the status of HPV integration makes any difference in the progression of cervical cancer. The purpose of the research is to reduce the miss of cervix lesions and prove that HPV integration detection is sensitive in cervical cancer precise screening.

SUMMARY:
The stratified analysis by the level of HPV DNA integration in HSIL and cervical cancer will be drawn to explore whether the status of HPV integration makes any difference in the progression of cervical cancer. The purpose of the research is to reduce the miss of cervix lesions and prove that HPV integration detection is sensitive in cervical cancer precise screening.

ELIGIBILITY:
Inclusion Criteria:

* HPV-positive patients； Patients have completed HPV detection, TCT, and HPV integration detection before surgery or biopsy； Patients with priced diagnoses accepted treatment according to ASCCP Risk-Based Management Consensus Guidelines for Abnormal Cervical Cancer Screening Tests and Cancer Precursors； Patients who are voluntary participants in this research and cooperate to follow-up with subscribing informed consent.

Exclusion Criteria:

* Patients who are not suitable for the trial； Patients existing other subtype malignancy tumors are still in treatment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is expected to be included in 2000 female in this study.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Tissue pathological diagnosis | 1year since HPV integrated test
  Tissue pathological diagnosis in 1 year since HPV integrated test

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Li, Principal Investigator — Tongji Hospital, Affiliated to Tongji Medical College of Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No